CLINICAL TRIAL: NCT02430311
Title: A Phase I, Open Label, 2 Part Study to Determine the Pharmacokinetics of Olaparib 300 mg bd Administered as Monotherapy and Olaparib 100 mg bd as Monotherapy and in Combination With Paclitaxel in Chinese Patients With Advanced Solid Tumours
Brief Title: The Pharmacokinetics and Safety of Olaparib Alone and With Paclitaxel in Chinese Patients With Advanced Solid Tumour.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D081BC00002
Record Dates: First submitted 2015-04-07; First posted 2015-04-30 (Estimated); Results first posted 2018-09-13 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Advanced Solid Tumours
Keywords: Chinese Patients
MeSH Terms: interventions — olaparib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Treat 15 patients, single dose olaparib 300mg followed by multiple dose olaparib 300mg twice a day
  Interventions: Drug: Olaparib
- Cohort 2 (Experimental): Treat 15 patients, single dose olaparib 100mg followed by multiple dose olaparib 100 mg twice a day and then in combination with paclitaxel (80mg/m2 weekly on days 1, 8 and 15 of a single 28-day cycle)
  Interventions: Drug: Paclitaxel; Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Tablet-150mg, Oral
  Arms: Cohort 1
Drug: Paclitaxel — Injection
  Arms: Cohort 2
Drug: Olaparib — Tablet-100mg, Oral
  Arms: Cohort 2

SUMMARY:
This is a 2 parts phase I, open label trial of olaparib monotherapy and olaparib in combination with paclitaxel in patients with solid tumours. Part A will assess the single and multiple dose pharmacokinetics of olaparib monotherapy and multiple dose pharmacokinetics of olaparib in combination with paclitaxel. Part B will assess the safety of multiple doses of olaparib in Cohort 1 and of olaparib when co-administered with paclitaxel in Cohort 2

DETAILED DESCRIPTION:
Part A will access the pharmacokinetics of olaparib: Cohort 1 will investigate the single and multiple dose pharmacokinetics of olaparib following 300mg bd monotherapy dose(s); Cohort 2 will investigate the single and multiple dose pharmacokinetics of olaparib following 100mg bd monotherapy dose(s) and the multiple dose pharmacokinetics in the presence of co-administered paclitaxel (80mg/m2 weekly on days 1, 8 and 15 of a single 28-day cycle).

In Part B: Safety profile of olaparib 300mg bd as monotherapy and olaparib 100mg bd in combination with weekly paclitaxel will also be investigated in Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent
2. Patient aged ≥ 18 years
3. Histologically or, where appropriate, cytologically confirmed malignant solid tumour refractory or resistant to standard therapy and for which no suitable effective standard therapy exists
4. life expectancy of ≥ 12 weeks
5. Patients for Cohort 2 must be eligible for paclitaxel treatment
6. Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations
7. ECOG performance status ≤ 2
8. Satisfactory organ and bone marrow function measured within 28 days prior to administration of study treatment including - Haemoglobin ≥ 10.0 g/dL and no blood transfusion in the 4 weeks prior to the first dosing of study drug. - Absolute neutrophil count ≥ 1.5 × 109/L
9. Evidence of non-childbearing status for women of childbearing potential, or postmenopausal status: negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on Day 1.
10. Patients must be on a stable concomitant medication regimen, defined as no changes in medication or in dose within 2 weeks prior to start of olaparib dosing, except for bisphosphonates, denosumab and corticosteroids, which should be stable for at least 4 weeks prior to start of olaparib dosing.

Exclusion criteria:

1. Involvement in the planning and/or conduct of the study.
2. Previous enrolment in the present study.
3. Treatment with any investigational product during the last 14 days (or a longer period depending on the defined characteristics of the agents used).
4. Any previous treatment with a Poly (ADP-ribose) polymerase (PARP) inhibitor, including olaparib.
5. Patients with other malignancy within the last 5 years, except adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, ductal carcinoma in situ, Stage 1, Grade 1 endometrial cancer, or other solid tumours including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥5 years.
6. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication. These include patients with gastric or intestinal cancer or patients with prior surgical procedures such as full or partial gastrectomy.
7. Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 4 weeks from the last dose prior to study treatment.
8. Concomitant use of known potent CYP3A4 (Cytochrome P450 3A4) inhibitors.
9. Patients with any ongoing toxicities (>CTCAE (Common Terminology Criteria for Adverse Events) grade 2), with the exception of alopecia, caused by previous cancer therapy.
10. Resting ECG with QTc (Heart Rate Corrected QT interval) > 470msec or family history of long QT syndrome.
11. Patients with interstitial pneumonia or diffused symptomatic fibrosis of the lungs.
12. Patients with myelodysplastic syndrome/acute myeloid leukaemia.
13. Patients with symptomatic uncontrolled brain metastases.
14. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
15. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection.
16. Immunocompromised patients, e.g. patients who are known to be serologically positive for human immunodeficiency virus (HIV).
17. Patients with known active hepatic disease (i.e. Hepatitis B or C).
18. Patients with a known hypersensitivity to olaparib, paclitaxel or any of the excipients of the product.
19. Breastfeeding women.
20. Clinical judgement by the investigator that the patient should not participate in the study.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2016-07-27 (Actual); Study Completion 2017-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, MD, Principal Investigator — Cancer Institute and Hospital (CIH), Chinese Academy of Medical Sciences and Peking Union Medical College; Jianming Xu, MD, Principal Investigator — 307 Hospital of Military Medical Sciences; Jianzhong Shentu, Principal Investigator — No.1 Affiliated Hospital of College of Medicine, Zhejiang University
Locations (2):
- China (2):
  - Research Site, Beijing
  - Research Site, Hangzhou

REFERENCES:
- [Background] Yuan P, Shentu J, Xu J, Burke W, Hsu K, Learoyd M, Zhu M, Xu B. Pharmacokinetics and safety of olaparib tablets as monotherapy and in combination with paclitaxel: results of a Phase I study in Chinese patients with advanced solid tumours. Cancer Chemother Pharmacol. 2019 May;83(5):963-974. doi: 10.1007/s00280-019-03799-1. Epub 2019 Mar 18. PMID 30887180
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081BC00002&attachmentIdentifier=b60a2fb8-5bbd-446e-a489-b69d309fdbca&fileName=CSP_Final_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was performed at 3 study centres in China.The first patient entered the study on 10 June 2015 and the last patient completed Part A of the study on 02 August 2016, and the date of last patient last visit in Part B was 28 April 2017.
Pre-assignment Details: 47 patients were screened in the study. 11 patients were not assigned to treatment due to eligibility criteria not fulfilled. 5 patients excluded from the PK analysis set due to previous gastric surgery. 1 of the 5 patients was also excluded due to vomiting within 3 hours of dosing on a PK day or on the 3 days prior to a multiple dose PK Day.
Groups:
- Cohort 1: Olaparib 300 mg alone
- Cohort 2: Olaparib 100 mg bd in combination with paclitaxel
Period: Part A
Arm/Group | Cohort 1 | Cohort 2
Started | 20 | 16
Received Olaparib | 20 | 16
Received Paclitaxel | 0 (Cohort 1 patients are planned to receive olaparib monotherapy) | 16
Completed | 19 | 15
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Part B
Arm/Group | Cohort 1 | Cohort 2
Started | 19 | 15
Received Olaparib | 19 | 15
Received Paclitaxel | 0 (Cohort 1 patients are planned to receive olaparib monotherapy) | 14
Completed | 9 | 7
Not Completed | 10 | 8
Not completed — Meet study-specific withdrawal criteria | 6 | 6
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 20 | 16 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (10.43) | 49.3 (9.49) | 48.4 (9.92)
Age, Customized [Number; unit: Participants]
  <50 years | 11 | 9 | 20
  ≥50 <65 years | 9 | 6 | 15
  ≥65 <75 years | 0 | 1 | 1
  ≥75 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 7 | 1 | 8
Race/Ethnicity, Customized [Number; unit: Participants]
  Chinese | 20 | 16 | 36
Height [Mean (Standard Deviation); unit: cm] | 164.9 (6.25) | 160.3 (4.81) | 162.8 (6.04)
Weight [Mean (Standard Deviation); unit: kg] | 64.8 (10.35) | 60.9 (8.71) | 63.1 (9.71)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 23.91 (4.144) | 23.78 (3.599) | 23.85 (3.857)

OUTCOME MEASURES:

1. Primary Outcome: Single Dose PK Parameter--Cmax
Description: Single dose PK parameter summary for olaparib in monotherapy by dose - Cmax (PK analysis set)
Time Frame: PK samples were collected pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 (Day 2) and 48 h (Day 3)
Population: PK analysis set, which includes all patients who receive an olaparib dose and provide evaluable PK profiles in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 16 | 15
µg/mL | 6.875 (39.70) | 2.972 (41.80)

2. Primary Outcome: Single Dose PK Parameter--AUC
Description: Single dose PK parameter summary for olaparib in monotherapy by dose - AUC (PK analysis set)
Time Frame: PK samples were collected pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 (Day 2) and 48 h (Day 3)
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 16 | 15
µg*h/mL
  AUC0-12 | 31.68 (52.97) | 10.86 (61.60)
  AUC0-t | 36.37 (59.58) | 12.63 (75.42)
  AUC | 36.53 (59.86) | 12.75 (76.70)

3. Primary Outcome: Single Dose PK Parameter--tmax
Description: Single dose PK parameter summary for olaparib in monotherapy by dose - tmax (PK analysis set)
Time Frame: PK samples were collected pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 (Day 2) and 48 h (Day 3)
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 2 | Cohort 1
Number analyzed (Participants) | 15 | 16
hour | 1.95 (61.60) [0.98 to 4.00] | 1.50 [0.50 to 4.00]

4. Primary Outcome: Single Dose PK Parameter--t1/2, λz
Description: Single dose PK parameter summary for olaparib in monotherapy by dose - t1/2, λz (PK analysis set)
Time Frame: PK samples were collected pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 (Day 2) and 48 h (Day 3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cohort 2 | Cohort 1
Number analyzed (Participants) | 15 | 16
hour | 7.165 (2.542) [3.60 to 11.5] | 6.519 (1.346) [4.62 to 8.82]

5. Primary Outcome: Single Dose PK Parameter--Vz/F
Description: Single dose PK parameter summary for olaparib in monotherapy by dose - Vz/F (PK analysis set)
Time Frame: PK samples were collected pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 (Day 2) and 48 h (Day 3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Cohort 2 | Cohort 1
Number analyzed (Participants) | 15 | 16
L | 88.32 (44.04) [3.60 to 11.5] | 74.78 (75.41)

6. Primary Outcome: Single Dose PK Parameter--CL/F
Description: Single dose PK parameter summary for olaparib in monotherapy by dose - CL/F (PK analysis set)
Time Frame: PK samples were collected pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 (Day 2) and 48 h (Day 3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort 2 | Cohort 1
Number analyzed (Participants) | 15 | 16
L/h | 9.217 (4.531) [3.60 to 11.5] | 8.107 (6.689)

7. Primary Outcome: Steady State PK Parameter--Cmax, ss and Cmin, ss at Day 8
Description: Steady state pharmacokinetic parameter summary for olaparib by dose and visit after multiple doses - Cmax, ss and Cmin, ss (PK analysis set)
Time Frame: PK samples were collected pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 h post morning dose of Day 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Cohort 2 (Olaparib Alone): Cohort 2 patients with olaparib 100 mg alone dosed
Arm/Group | Cohort 1 | Cohort 2 (Olaparib Alone)
Number analyzed (Participants) | 15 | 15
µg/mL
  Cmax, ss | 8.268 (35.02) | 3.752 (40.99)
  Cmin, ss | 0.7996 (117.8) | 0.3162 (129.4)

8. Primary Outcome: Steady State PK Parameter--AUCss at Day 8
Description: Steady state pharmacokinetic parameter summary for olaparib by dose and visit after multiple doses - AUC (PK analysis set)
Time Frame: PK samples were collected pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 h post morning dose of Day 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Groups:
- Cohort 2, Olaparib Alone: Cohort 2 patients with olaparib 100 mg alone dosed
Arm/Group | Cohort 1 | Cohort 2, Olaparib Alone
Number analyzed (Participants) | 15 | 15
µg*h/mL
  AUCss | 43.95 (48.43) | 16.73 (61.38)
  AUC0-t | 43.91 (48.47) | 16.68 (61.30)

9. Primary Outcome: Steady State PK Parameter--tmax, ss at Day 8
Description: Steady state pharmacokinetic parameter summary for olaparib by dose and visit after multiple doses - tmax, ss (PK analysis set)
Time Frame: PK samples were collected pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 h post morning dose of Day 8
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1 | Cohort 2, Olaparib Alone
Number analyzed (Participants) | 15 | 15
hour | 1.50 [0.97 to 3.00] | 2.00 [0.97 to 4.02]

10. Primary Outcome: Steady State PK Parameter--RAC and TCP at Day 8
Description: Steady state pharmacokinetic parameter summary for olaparib by dose and visit after multiple doses - RAC and TCP (PK analysis set)
Time Frame: PK samples were collected pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 h post morning dose of Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1 | Cohort 2, Olaparib Alone
Number analyzed (Participants) | 15 | 15
Ratio
  RAC | 1.436 (0.2081) | 1.565 (0.2984)
  TCP | 1.253 (0.2150) | 1.349 (0.3349)

11. Primary Outcome: Steady State PK Parameter--Cmax, ss and Cmin, ss at Day 9
Description: as for outcome 7
Time Frame: PK samples were collected pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 h post morning dose of Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Cohort 2(Olaparib 100 mg + Paclitaxel): Cohort 2 patients with Olaparib 100 mg dosed in combination with paclitaxel
Arm/Group | Cohort 2(Olaparib 100 mg + Paclitaxel)
Number analyzed (Participants) | 15
µg/mL
  Cmax, ss | 3.031 (56.14)
  Cmin, ss | 0.1915 (125.2)

12. Primary Outcome: Steady State PK Parameter--AUCss at Day 9
Description: as for outcome 8
Time Frame: PK samples were collected pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 h post morning dose of Day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Cohort 2(Olaparib 100 mg + Paclitaxel)
Number analyzed (Participants) | 15
µg*h/mL
  AUCss | 12.44 (57.46)
  AUC0-t | 12.42 (57.36)

13. Primary Outcome: Steady State PK Parameter--tmax, ss at Day 9
Description: as for outcome 9
Time Frame: PK samples were collected pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 h post morning dose of Day 9
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 2(Olaparib 100 mg + Paclitaxel)
Number analyzed (Participants) | 15
hour | 1.48 (61.38) [0.28 to 5.95]

14. Primary Outcome: Steady State PK Parameter--CLss/F at Day 8
Description: Steady state pharmacokinetic parameter summary for olaparib by dose and visit after multiple doses - CLss/F (PK analysis set)
Time Frame: PK samples were collected pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 h post morning dose of Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort 1 | Cohort 2, Olaparib Alone
Number analyzed (Participants) | 15 | 15
L/h | 7.512 (3.418) | 6.745 (2.923)

ADVERSE EVENTS:
Time Frame: Includes AEs with an onset date between the first dose date in the appropriate Part and the day before first dose in Part B (for Part A only), or 30 days following the date of last dose of study medication if the subject discontinued.
Groups:
- Cohort 1 Part A: Part A Olaparib 300 mg alone
- Cohort 2 Part A, Olaparib 100 mg: Part A Cohort 2 patients, who have received olaparib 100 mg monotherapy treatment
- Cohort 2 Part A, Olaparib 100mg in Combination With Paclitaxel: Part A Cohort 2 patients, who have received olaparib 100 mg + paclitaxel treatment
- Cohort 1 Part B: Part B Olaparib 300 mg alone
- Cohort 2 Part B, Olaparib 300 mg Monotherapy: Part B Cohort 2 patients, who continued on Olaparib 300mg monotherapy after completed combination therapy
- Cohort 2 Part B, Olaparib 100mg in Combination With Paclitaxel: Part B Cohort 2 patients, who have received olaparib 100 mg + paclitaxel treatment
Arm/Group | Cohort 1 Part A | Cohort 2 Part A, Olaparib 100 mg | Cohort 2 Part A, Olaparib 100mg in Combination With Paclitaxel | Cohort 1 Part B | Cohort 2 Part B, Olaparib 300 mg Monotherapy | Cohort 2 Part B, Olaparib 100mg in Combination With Paclitaxel
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/16 | 4/16 | 0/19 | 0/2 | 1/15
Other Adverse Events (participants affected / at risk) | 11/20 | 8/16 | 16/16 | 18/19 | 2/2 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Part A (N=20) | Cohort 2 Part A, Olaparib 100 mg (N=16) | Cohort 2 Part A, Olaparib 100mg in Combination With Paclitaxel (N=16) | Cohort 1 Part B (N=19) | Cohort 2 Part B, Olaparib 300 mg Monotherapy (N=2) | Cohort 2 Part B, Olaparib 100mg in Combination With Paclitaxel (N=15)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Part A (N=20) | Cohort 2 Part A, Olaparib 100 mg (N=16) | Cohort 2 Part A, Olaparib 100mg in Combination With Paclitaxel (N=16) | Cohort 1 Part B (N=19) | Cohort 2 Part B, Olaparib 300 mg Monotherapy (N=2) | Cohort 2 Part B, Olaparib 100mg in Combination With Paclitaxel (N=15)
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 8
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 2 | 5 | 4 | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2 | 2 | 3 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1
Faeces hard (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 9 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0 | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 8 | 5 | 0 | 2
Asthenia (General disorders) | 0 | 1 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 1 | 0 | 2
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2 | 3 | 0 | 4
Alanine aminotransferase increased (Investigations) | 0 | 1 | 3 | 4 | 0 | 5
Weight decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 2 | 1 | 0 | 1
Blood albumin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 2 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 1 | 12 | 8 | 1 | 15
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 11 | 8 | 1 | 14
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 6 | 7 | 1 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1 | 1 | 2 | 0 | 1
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 3 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 2
Axillary pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Protein urine present (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Poor quality sleep (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Xerophthalmia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Principal Investigator may use the Study results (data generated at the site) and shall not publish or present any such results until the earlier of (i) the date of the first Study results publication and (ii) the end of the eighteen (18) month period following the completion, or early termination, of the Study at all participating sites.